CLINICAL TRIAL: NCT00104182
Title: Efficacy and Safety Comparison of Insulin Detemir Morning, Insulin Detemir Evening and NPH Insulin Evening as Add-on to Oral Antidiabetic Drug(s) in Patients With Type 2 Diabetes
Brief Title: Comparison of Insulin Detemir Morning, Insulin Detemir Evening and NPH Insulin Evening in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1632; 2004-001461-18 (EudraCT Number)
Record Dates: First submitted 2005-02-23; First posted 2005-02-24 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this trial is to compare the use of Insulin Detemir once a day (morning or evening) to NPH Insulin once a day (evening) when added to treatment with oral antidiabetic drugs in patients with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 months
* Currently treated with Oral Antidiabetic Drugs
* BMI lesser than or equal to 40 kg/m2
* HbA1c greater than or equal 7.5 and lesser than or equal to 11%

Exclusion Criteria:

* Proliferative retinopathy or maculopathy
* Recurrent major hypoglycaemia
* uncontrolled hypertension or any disease or condition (such as renal, hepatic or cardiac) that according to the judgement of the Investigator makes the subject unsuitable for participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2005-02; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
HbA1C | after 20 weeks

SECONDARY OUTCOMES:
Adverse events
body weight
Hypoglycemia
Blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (91):
- United States (29):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Fall River, Massachusetts
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Lewiston, New York
  - Novo Nordisk Investigational Site, Williamsville, New York
  - Novo Nordisk Investigational Site, Grand Forks, North Dakota
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Connellsville, Pennsylvania
  - Novo Nordisk Investigational Site, Lancaster, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Conroe, Texas
  - Novo Nordisk Investigational Site, Killeen, Texas
  - Novo Nordisk Investigational Site, Seattle, Washington
- Denmark (12):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Glostrup Municipality
  - Novo Nordisk Investigational Site, Herlev
  - Novo Nordisk Investigational Site, Hillerød
  - Novo Nordisk Investigational Site, Hjørring
  - Novo Nordisk Investigational Site, Horsens
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, København S
  - Novo Nordisk Investigational Site, Næstved
  - Novo Nordisk Investigational Site, Roskilde
- France (10):
  - Novo Nordisk Investigational Site, Bagnols-sur-Cèze
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Carcassonne
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, Dax
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Quimper
  - Novo Nordisk Investigational Site, Rueil-Malmaison
  - Novo Nordisk Investigational Site, Tours
  - Novo Nordisk Investigational Site, Vénissieux
- Italy (12):
  - Novo Nordisk Investigational Site, Cagliari
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Genova
  - Novo Nordisk Investigational Site, Messina
  - Novo Nordisk Investigational Site, Monza
  - Novo Nordisk Investigational Site, Napoli
  - Novo Nordisk Investigational Site, Parma
  - Novo Nordisk Investigational Site, Pescara
  - Novo Nordisk Investigational Site, Prato
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Torino
  - Novo Nordisk Investigational Site, Treviso
- Netherlands (7):
  - Novo Nordisk Investigational Site, 's-Hertogenbosch
  - Novo Nordisk Investigational Site, Almelo
  - Novo Nordisk Investigational Site, Etten-Leur
  - Novo Nordisk Investigational Site, Roelofarendsveen
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Vlodrop
- Norway (7):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Elverum
  - Novo Nordisk Investigational Site, Gjøvik
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- Spain (14):
  - Novo Nordisk Investigational Site, Alcorcón
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Bilbao
  - Novo Nordisk Investigational Site, Cadiz
  - Novo Nordisk Investigational Site, Getafe
  - Novo Nordisk Investigational Site, Gijón
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Pamplona
  - Novo Nordisk Investigational Site, Santa Cruz de Tenerife
  - Novo Nordisk Investigational Site, Santiago de Compostela
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Valladolid

REFERENCES:
- [Result] Philis-Tsimikas A, Charpentier G, Clauson P, Ravn GM, Roberts VL, Thorsteinsson B. Comparison of once-daily insulin detemir with NPH insulin added to a regimen of oral antidiabetic drugs in poorly controlled type 2 diabetes. Clin Ther. 2006 Oct;28(10):1569-81. doi: 10.1016/j.clinthera.2006.10.020. PMID 17157113
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com